CLINICAL TRIAL: NCT03882996
Title: Long-Term, Open-Label, Safety and Tolerability Study of Ezetimibe (SCH 58235) in Addition to Atorvastatin in Subjects With Coronary Heart Disease or Multiple Risk Factors and With Primary Hypercholesterolemia Not Controlled by a Starting Dose (10 mg) of Atorvastatin
Brief Title: A Long-term Safety and Tolerability Study of Ezetimibe Plus Atorvastatin in Participants With Coronary Heart Disease, Multiple Risk Factors, or Hypercholesterolemia Not Controlled by Atorvastatin (P01418/MK-0653-032)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01418; MK-0653-032 (Other: Merck); P01418 (Other: Merck)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezetimibe 10 mg + Atorvastatin (Experimental): Ezetimibe 10 mg plus atorvastatin 10 to 80 mg daily for up to 12 months
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg daily in the morning
  Other Names: Zetia®; SCH 058235; MK-0653
Drug: Atorvastatin — Atorvastatin 10 mg daily in the morning. Atorvastatin dose could be titrated up (by doubling the dose up to a maximum of 80 mg daily) to achieve the target low-density-lipoprotein cholesterol (LDL-C) level of 100 mg/dL (2.59 mmol/L) after a minimum of 4 weeks of treatment.
  Other Names: Lipitor®; SCH 412387; MK-9396

SUMMARY:
The purpose of this study was to evaluate the long-term safety and tolerability of ezetimibe 10 mg once daily co-administered with atorvastatin 10 to 80 mg daily for up to 12 consecutive months in participants with heterozygous familial hypercholesterolemia (HeFH) or in participants with coronary heart disease (CHD) or multiple cardiovascular risk factors and primary hypercholesterolemia not controlled by a starting dose (10 mg daily) of atorvastatin.

DETAILED DESCRIPTION:
Adult participants with a diagnosis of HeFH or CHD or multiple risk factors (≥2) and with primary hypercholesterolemia who had successfully completed the 14-week, double-blind efficacy and safety study of ezetimibe co-administered with atorvastatin (Protocol No. P00693/MK-0653-030; NCT03867318) were eligible for enrollment in this long-term extension study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have successfully completed the 14-week double-blind, efficacy and safety study of SCH 58235 in addition to atorvastatin in participants with CHD or multiple risk factors or HeFH, (Protocol P00693/MK-0653-030; NCT03867318). Entry into this protocol must occur at the time of completion of Protocol P00693/MK-0653-030; NCT03867318
* All women must have a negative pregnancy test prior to study entry. Women of child bearing potential must agree to practice an effective barrier method of birth control for the duration of the study. In addition, participants must agree to practice an effective barrier method of birth control for 30 days following the last dose of atorvastatin administered
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable estrogen (ERT), estrogen/progestin (HRT) or raloxifene regimen during study period

Exclusion Criteria:

* Participants who discontinued from the Protocol P00693 due to adverse events or poor compliance
* Pregnant or lactating women
* Participants who are known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2000-10-06 (Actual); Primary Completion 2003-02-04 (Actual); Study Completion 2003-02-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced an adverse event | Up to 12 months
Number of participants who discontinued study drug due to an adverse event | Up to 12 months

SECONDARY OUTCOMES:
Percentage of participants achieving target LDL-C level (≤100 mg/dL) | Up to 12 months
Change from baseline in LDL-C levels | Up to 12 months
Change from baseline in HDL-C levels | Up to 12 months
Change from baseline in triglyceride levels | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC